CLINICAL TRIAL: NCT00371579
Title: Treatment With Rosuvastatin in Patients With Hepatitis C
Brief Title: Rosuvastatin for Hepatitis C
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no actual patients recruited within year 1 after ethical committee approval
Sponsor: UMC Utrecht (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06-125
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2009-02

CONDITIONS: Hepatitis C
Keywords: rosuvastatin; hepatitis C; geranylgeranylation; HCV-RNA load
MeSH Terms: conditions — Hepatitis C | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: rosuvastatin

SUMMARY:
Objective: Determine if maximum doses of rosuvastatin are safe in patients infected with hepatitis C and if the so called pleiotropic effects of rosuvastatin cause a decrease in the HCV viral load.

Primary study parameters: 1. to which extend causes rosuvastatin serious side effects like rhabdomyolysis and hepatotoxicity in patients chronically infected with hepatitis C? 2. does treatment with rosuvastatin in HCV infected patients lead to lower HCV-RNA viral load? 3. Is a decrease in LDL correlated to a decrease in HCV-RNA load?

DETAILED DESCRIPTION:
Study design: it's a pilot study in which the patients form their own control group. A total of 10 patients will be included. To evaluate the effect of maximum doses of rosuvastatin on liver function and side effects, first 2 patients will be treated and evaluated. If they experience no serious adverse events then a further 8 patients will be included. The dose of rosuvastatin will be increased over a period of 4 weeks.

Intervention: based on experience in treating dyslipidemia, gradually increasing the dose of rosuvastatin diminishes the experienced side effects and decreases the chances of developing hepatotoxicity. Therefore in this study we chose to increase the dose (see flowchart). Patients will start with 5 mg a day wich will be increased after 1 week to 10 mg per day. After the second week of therapy a further increase to 20 mg per day is executed. This dose will be given for another 2 weeks. At week 4 of treatment a further increase to 40 mg is done.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* All patients with hepatitis C (all genotypes)
* negative for hepatitis B and HIV
* ALAT < 2,5 x below the upper limit of normal
* serological evidence of hepatitis C infection with detectable HCV-RNA (with Bayer Versant HCV bDNA V3.0)
* failed current standard of care treatment with peginterferon and ribavirin
* WHO-score ≤1
* fertile women must have a negative pregnancy test in the week before start of medication. Use of contraceptives during the whole study-period
* physically and mentally able to attend outpatients clinics

Exclusion Criteria:

* Hepatitis C patiënts naive for (peg)interferon and ribavirin treatment
* Alcohol abuses (> 20 grams per day) in the last year
* liver cirrhosis detected through liver biopsy or decompensated liver disease (child-pugh B or C)
* concomitant treatment with hepatotoxic medication / interfering with CYP450 system: anti-fungal medication (voriconazole), antibiotics (gentamycine, azitromycine, claritromycin, erytromycin), immuun-suppresive drugs (cyclosporine), anti-arythmia (diltiazem, verapamil) and tuberculostatic drugs (rifampicin).
* current statin use
* active pregnancy or wish of pregnangy
* use of grapefruit juice
* mentally not fit to participate in the study
* daily use of more than 2 grams of paracetamol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
occurrence of serious side effects like rhabdomyolysis and hepatotoxicity during treatment
decrease of HCV-RNA viral load during treatment
decrease of LDL during treatment

CONTACTS AND LOCATIONS:
Overall Officials: I.M. Hoepelman, Professor, Principal Investigator — UMC Utrecht; H. Lokhorst, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Kapadia SB, Chisari FV. Hepatitis C virus RNA replication is regulated by host geranylgeranylation and fatty acids. Proc Natl Acad Sci U S A. 2005 Feb 15;102(7):2561-6. doi: 10.1073/pnas.0409834102. Epub 2005 Feb 7. PMID 15699349
- [Background] Ye J, Wang C, Sumpter R Jr, Brown MS, Goldstein JL, Gale M Jr. Disruption of hepatitis C virus RNA replication through inhibition of host protein geranylgeranylation. Proc Natl Acad Sci U S A. 2003 Dec 23;100(26):15865-70. doi: 10.1073/pnas.2237238100. Epub 2003 Dec 10. PMID 14668447